CLINICAL TRIAL: NCT01047046
Title: Use of Combined Anticholinergic Medication and Sacral Neuromodulation in the Treatment of Refractory Overactive Bladder
Brief Title: Combined Anticholinergic Medication and Sacral Neuromodulation to Treat Refractory Overactive Bladder
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Karen Noblett, MD, UC Irvine Medical Center
Other Study IDs: 2008-6162
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Last update posted 2010-07-15 (Estimated); Status verified 2010-07

CONDITIONS: Overactive Bladder
Keywords: SNM device; Chart review of patients with surgical placed SNM device
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- SNM device placement: Patients who have undergone a placement of a SNM device to treat refractory OAB. A retrospective chart review will be performed on all patients who underwent a one or two-stage placement of an SNM device, which includes an implantable pulse generator (IPG), for refractory urge incontinence and urgency frequency symptoms. The patients will be those of Dr. Karen Noblett, having their device placed after 2001.
  Interventions: Other: Retrospective chart review

INTERVENTIONS:
Other: Retrospective chart review — This study is a retrospective chart review including all patients who received surgical placement of a SNM device with Dr. Noblett from 2001 to the present.
  The following data will be collected from patient charts: age at time of surgery, gravidity/parity, body mass index, pre-existing medical conditions/surgical history, current medications, menopausal status, form and severity of OAB symptoms, other previously or currently used interventions, method of SNM device placement, observed motor/sensory response, percent improvement of symptoms, follow-up OAB symptoms, frequency of InterStim settings adjustments, adverse events, significant changes in health, and incidence/reason for drop out.

SUMMARY:
This study is a retrospective chart review including all patients who received surgical placement of a SNM device with Dr. Noblett from 2001 to the present.

DETAILED DESCRIPTION:
The following data will be collected from patient charts: age at time of surgery, gravidity/parity, body mass index, pre-existing medical conditions/surgical history, current medications, menopausal status, form and severity of OAB symptoms, other previously or currently used interventions, method of SNM device placement, observed motor/sensory response, percent improvement of symptoms, follow-up OAB symptoms, frequency of InterStim settings adjustments, adverse events, significant changes in health, and incidence/reason for drop out.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with symptoms of OAB, namely urge incontinence and urgency-frequency.
* Ages 18 and older.

Exclusion Criteria:

* Any patient who received surgical placement of an SNM device to treat non-obstructive urinary retention, or the symptoms of an underlying neurologic pathology, such as Parkinson's or Multiple Sclerosis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone a placement of a SNM device to treat refractory OAB. A retrospective chart review will be performed on all patients who underwent a one or two-stage placement of an SNM device, which includes an implantable pulse generator (IPG), for refractory urge incontinence and urgency frequency symptoms. The patients will be those of Dr. Karen Noblett, having their device placed after 2001.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of combined therapy - determine the nmbr of pts on anticholinergic medication to treat symptoms of OAB after placement of SNM device, examine outcomes and defining characteristics of these pts compared to those not receiving anticholinergics. | Retrospective chart review

SECONDARY OUTCOMES:
Predictors of SNM therapy success - collect data factors; previously trialed conservative therapies, age, and severity of urinary symptoms, and examine for a correlation with urinary symptom resolution with either SNM therapy or combined therapy. | Retrospective chart review

CONTACTS AND LOCATIONS:
Overall Officials: Karen Noblett, MD, Principal Investigator — UCI Medical Center
Locations (1):
- UCI Women's Healthcare, Orange, California, United States